CLINICAL TRIAL: NCT04526236
Title: Influence of Aging on Perioperative Methadone Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190510001
Record Dates: First submitted 2020-08-05; First posted 2020-08-25 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative; Opioid Use; Methadone Overdose of Undetermined Intent
Keywords: Methadone; Elderly; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into four groups according to the dose of intravenous methadone to be administered during anesthetic induction, for a total number of 60 patients.
Who Masked: Participant, Care Provider
Masking Description: The masking will be generated on a research laboratory computer and will be stored in an encrypted file. This information will be known exclusively to a member of the research team present during the surgery, who will hand over preparing the corresponding medicine in a 20 cc syringe and hand it over to the treating anesthesiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Methadone 0 (Placebo Comparator): Induction will be performed with a bolus of propofol, continuous infusion of remifentanil, and rocuronium. Once the patient is intubated and has hemodynamic stability will be administered the placebo drug.
  Interventions: Drug: Methadone Injectable Product
- Methadone 1 (Experimental): Induction will be performed with a bolus of propofol, continuous infusion of remifentanil, and rocuronium. Once the patient is intubated and has hemodynamic stability will be administered an intravenous methadone dose of 0.05 mg/kg.
  Interventions: Drug: Methadone Injectable Product
- Methadone 2 (Experimental): Induction will be performed with a bolus of propofol, continuous infusion of remifentanil, and rocuronium. Once the patient is intubated and has hemodynamic stability will be administered an intravenous methadone dose of 0.1 mg/kg.
  Interventions: Drug: Methadone Injectable Product
- Methadone 3 (Experimental): Induction will be performed with a bolus of propofol, continuous infusion of remifentanil, and rocuronium. Once the patient is intubated and has hemodynamic stability will be administered an intravenous methadone dose of 0.2 mg/kg.
  Interventions: Drug: Methadone Injectable Product

INTERVENTIONS:
Drug: Methadone Injectable Product — Perioperative use of placebo for pain management and remifentanil during the surgery.
  Other Names: Methadone 0; Methadone 1 0,05 mg/kg; Methadone 2 0,1 mg/kg; Methadone 3 0,2 mg/kg

SUMMARY:
Increasingly, elderly patients undergo anesthesia and surgery. Methadone is a great opioid for perioperative pain management, however, to date there are no pharmacokinetic or pharmacodynamic studies that asses a methadone dose adjustment in the elderly patient. The present study is aimed to characterize the pharmacokinetic and pharmacodynamic age-related changes of methadone in the adult population and further to design reference dosing protocols for intraoperative methadone use according to patient age.

DETAILED DESCRIPTION:
The subjects will be recruited from adult patients who undergo elective laparoscopic abdominal surgery at UC Christus Clinical Hospital (Santiago, de Chile). Patients will be randomly divided into four groups according to the dose of intravenous methadone to be administered during anaesthetic induction.

BIS-guided and standard general anaesthesia will be administered with routine monitoring. Methadone will be administered once the patient is intubated and has hemodynamic stability. The only opioids that patients will receive will be remifentanil and methadone.

Upon admission to the Post-anesthesia care unit, the patient is given a Patient-Control Analgesia pump for intravenous administration of morphine. Clinic evaluations will be carried out periodically and blood samples for measurement of plasma methadone will be taken at different times. Samples will be analyzed using high-performance liquid chromatography spectrofluorometric method. The data obtained will be collected in a form within the REDCAP application, to subsequently generate an encrypted database. Groups will be compared regarding pain score, drugs used, opioid consumption, side effects, time of recovery, and patient satisfaction.

One, two and three-compartment linear models will be used to fit the plasma methadone concentration data over time. Models are parameterized in terms of elimination clearance, compartment distribution clearance, central volume and peripheral volume of distribution, as appropriate. The use of rescue morphine in the Post-anesthesia care unit will be used as a measure to relate the methadone dose (mg/kg) with the analgesic efficacy using an EMAX model. The data will be modelled using NONMEM VII. A proportional term will be used for variability between subjects. Additive and proportional terms will be used to characterize the unknown residual variability.

Sample size calculations were estimated using a simulation-based approach and previous work with a similar methodology. To achieve an adequate representation of all age groups 60 patients will be required, distributed among 20 patients between 18 and 40 years, 20 patients between 41 and 65 years, and 20 patients> 65 years.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years.
2. ASA I, II or III.
3. Laparoscopic Abdominal Surgery.

Exclusion Criteria:

1. BMI> 35
2. Use of opioids up to 5 days before surgery.
3. Acute Liver Failure or Chronic Liver Damage Child C.
4. Kidney damage with creatinine clearance estimated by Cockcroft-Gault formula <60 ml/min.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Methadone plasmatic levels Measured by high pressure liquid chromatography | From the first dose up to 24 hours.
  Five venous blood samples will be taken from each patient for methadone plasmatic level analysis. Patients will be randomly divided into two groups with different sample collection times. Group 1 at 0.05, 0.75, 1.5, 6, 18 hours post drug administration and Group 2 at 0.25, 1, 3, 12 and 24 hours.

SECONDARY OUTCOMES:
Hemodynamics | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs. Then, from the entrance to the recovery room every 30 minutes up to 180 minutes.
  Non invasive systolic and diastolic blood pressure monitoring (mmHg).
Heart Rate | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs. Then, from the entrance to the recovery room every 30 minutes up to 180 minutes.
  Heart rate (bpm)
Pulse oximetry | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs. Then, from the entrance to the recovery room every 30 minutes up to 180 minutes.
  % oximetry saturation
BIS | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  Depth of anesthesia will be recorded with BIS monitor. From 60 - 40
Respiratory rate | Every 30 minutes. Since entering the recovery room up to 180 mins.
  bpm
Numeric Pain Rating Scale | Every 30 minutes. Since entering the recovery room up to 180 mins.
  Numeric Pain rating scale in rest and movement, from 0 (no pain) to 10 (maximum pain).
Nausea or vomiting | Every 30 minutes. Since entering the recovery room up to 180 mins.
  Presence of nausea or vomiting in the recovery room.
Sedation (Ramsay Scale) | Every 30 minutes. Since entering the recovery room up to 180 mins.
  Ramsay scale (1-6)
Respiratory depression | Every 30 minutes. Since entering the recovery room up to 180 mins.
  Presence of respiratory depression in the recovery room. (Respiratory rate less than 8 bpm requiring oxygen therapy).
Other opioids and pain management drugs used during recovery stay | Since the admission to the recovery room up to 2 hours.
  Name and total doses, including Morphine PCA.
Intestinal transit recovery | Since the admission to the recovery room up to 2 hours.
  Time to first flatus, fist bowel movement and stool. Presence of abdominal bloating.

OTHER OUTCOMES:
Body fat | Once, before the anesthetic induction in the operating toom.
  Body fat (kilograms) by body impedance analysis.
Level of satisfaction with pain management: 10-point scale | Since the admission to the recovery room up to 2 hours.
  10-point scale: very unsatisfied to very satisfied.
Lean Mass | Once, before the anesthetic induction in the operating toom.
  Lean mass (kilograms) by body impedance analysis.
Total water | Once, before the anesthetic induction in the operating toom.
  Total water (kilograms) by body impedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Elgueta, MD, Principal Investigator — Associate Professor
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Sadean MR, Glass PS. Pharmacokinetics in the elderly. Best Pract Res Clin Anaesthesiol. 2003 Jun;17(2):191-205. doi: 10.1016/s1521-6896(03)00002-8. PMID 12817914
- [Background] Shafer SL. The pharmacology of anesthetic drugs in elderly patients. Anesthesiol Clin North Am. 2000 Mar;18(1):1-29, v. doi: 10.1016/s0889-8537(05)70146-2. PMID 10934997
- [Background] Minto CF, Schnider TW, Egan TD, Youngs E, Lemmens HJ, Gambus PL, Billard V, Hoke JF, Moore KH, Hermann DJ, Muir KT, Mandema JW, Shafer SL. Influence of age and gender on the pharmacokinetics and pharmacodynamics of remifentanil. I. Model development. Anesthesiology. 1997 Jan;86(1):10-23. doi: 10.1097/00000542-199701000-00004. PMID 9009935
- [Background] Schnider TW, Minto CF, Shafer SL, Gambus PL, Andresen C, Goodale DB, Youngs EJ. The influence of age on propofol pharmacodynamics. Anesthesiology. 1999 Jun;90(6):1502-16. doi: 10.1097/00000542-199906000-00003. PMID 10360845
- [Background] Hilmer SN, McLachlan AJ, Le Couteur DG. Clinical pharmacology in the geriatric patient. Fundam Clin Pharmacol. 2007 Jun;21(3):217-30. doi: 10.1111/j.1472-8206.2007.00473.x. PMID 17521291
- [Background] Kaiko RF, Wallenstein SL, Rogers AG, Grabinski PY, Houde RW. Narcotics in the elderly. Med Clin North Am. 1982 Sep;66(5):1079-89. doi: 10.1016/s0025-7125(16)31383-9. No abstract available. PMID 7132470
- [Background] Singleton MA, Rosen JI, Fisher DM. Pharmacokinetics of fentanyl in the elderly. Br J Anaesth. 1988 May;60(6):619-22. doi: 10.1093/bja/60.6.619. PMID 3377944
- [Background] Scott JC, Ponganis KV, Stanski DR. EEG quantitation of narcotic effect: the comparative pharmacodynamics of fentanyl and alfentanil. Anesthesiology. 1985 Mar;62(3):234-41. doi: 10.1097/00000542-198503000-00005. PMID 3919613
- [Background] Gallagher R. Methadone: an effective, safe drug of first choice for pain management in frail older adults. Pain Med. 2009 Mar;10(2):319-26. doi: 10.1111/j.1526-4637.2008.00551.x. Epub 2009 Jan 16. PMID 19207240
- [Background] Lugo RA, Satterfield KL, Kern SE. Pharmacokinetics of methadone. J Pain Palliat Care Pharmacother. 2005;19(4):13-24. PMID 16431829
- [Background] Gagnon B, Almahrezi A, Schreier G. Methadone in the treatment of neuropathic pain. Pain Res Manag. 2003 Fall;8(3):149-54. doi: 10.1155/2003/236718. PMID 14657982

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT04526236/Prot_SAP_000.pdf